CLINICAL TRIAL: NCT01600677
Title: Determining the Impact of a Medication Delivery Unit on Medication Adherence Immediately Following Hospitalization of Adults With Common Cardiac Conditions
Brief Title: Determining the Impact of a Medication Delivery Unit on Medication Adherence of Adults With Common Cardiac Conditions
Acronym: EMMA-RCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated on 2/28/13, low enrollment; last participant med visit 5/13/13.
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Steven M Handler, MD, PhD, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0031272
Record Dates: First submitted 2012-05-14; First posted 2012-05-17 (Estimated); Results first posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Medication Adherence; Medication Nonadherence; Adverse Reaction to Drug
Keywords: Experimental; Computerized medication delivery unit
MeSH Terms: conditions — Medication Adherence; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computerized medication delivery unit (Experimental): Those hospitalized patients that meet all inclusion and exclusion criteria will be provided with an EMMA MDU for use in their homes for the 90-day period immediately following discharge.
  Interventions: Device: Computerized medication delivery unit
- Usual care (Active Comparator): Those hospitalized patients that meet all inclusion and exclusion criteria will receive medications from a dedicated pharmacy, but continue to make their medications in their usual way for the 90-day period immediately following discharge.
  Interventions: Other: Usual care

INTERVENTIONS:
Device: Computerized medication delivery unit — The patient's prescriptions and refills are packaged in standard-sized blister cards and loaded into EMMA units. EMMA identifies each medication automatically-no patient input is required. When activated by the patient, the medications are selected from the blister cards and released into the delivery tray. EMMA will remain in the patient's home for a period of 90 days immediately following hospitalization. After 90 days, the EMMA MDU will become available for the next eligible patient. This maximizes the number of patients that can benefit form the MDU, while addressing the transition period when medication-reconciliation problems are most common.
  Other Names: Electronic Medication Management Assistant (EMMA)
  Arms: Computerized medication delivery unit
Other: Usual care — Those hospitalized patients that meet all inclusion and exclusion criteria will receive medications from a dedicated pharmacy, but continue to make their medications in their usual way for the 90-day period immediately following discharge.
  Arms: Usual care

SUMMARY:
The research study is a randomized controlled trial (RCT). The primary endpoint is to compare medication adherence of adult patients recently hospitalized with a diagnosis of common cardiac conditions who require medication assistance either by receiving usual care or by using a medication delivery unit. The overall study will last a total of 12 months. Each subject will be enrolled for a period of 90 days.

DETAILED DESCRIPTION:
Care transition interventions have been successful in reducing medication-related problems and associated rehospitalization primarily by focusing on medication reconciliation conducted by trained healthcare professionals. Programs to improve the medication reconciliation process have largely been effective but have limitations, including: the expenses associated with recruiting, training, and retaining care transition healthcare professionals; the ability to provide services within a finite geographic area; and the retrospective nature of the reconciliation process, which usually occurs in the home following hospital discharge.

Our short-term objective is to determine the impact of the INRange Systems Electronic Medication Management Assistant (EMMA) medication delivery unit (MDU) for adults that require medication assistance in their home immediately following an acute hospitalization with a diagnosis of a common cardiac condition. As part of this study, we will determine: (1) Medication adherence rates (# doses/doses scheduled; EMMA (intervention) vs. determined by manual monthly pill counts at days 1, 45 and 90 (control)); (2) Health service utilization; (3) Health economic assessment from health plan and societal perspectives; (4) Medication administration errors; (5) Patient experience and satisfaction; (6) Medication reconciliation errors (using medication discrepancy tool); (7) 30-day readmission rates; and (8) Factors related to continued use of the EMMA MDU.

Study Overview and Design: The research study design associated with this proposal is a randomized controlled trial (RCT) design. The primary endpoint is to compare medication adherence of adult patients recently hospitalized with a diagnosis of congestive heart failure who require medication assistance either by receiving usual care (i.e., the control group; take medications as they had before hospitalization) or by using a medication delivery unit (i.e., the intervention group; take medications only from the device, which will always differ from the usual way in which medications were taken prior to hospitalization).

Study duration: The overall study will last a total of 12 months. Each subject will be enrolled for a period of 90 days regardless of unit of randomization (i.e., control/usual care vs. intervention).

Subject Recruitment: One-hundred and sixty patients > 18 years old who are admitted to UPMC Presbyterian Hospital will be considered as potential study participants. Records of these patients will be pre-screened within 24 hours of admittance using inclusion and exclusion criteria that can be assessed without direct patient contact.

Participants who pass the initial/exclusion criteria will be visited by the Research Assistant following agreement by the patient's attending physician. The Research Assistant will introduce the goals and design of the study, take informed consent, and complete the remaining exclusion instruments, MMSE, CAM, the test of the medication delivery unit interface, and questions regarding subjects' travel and hospice plans.

Detailed Description of Research Activities to be Performed: Following administrative medical record review by the UPMC Case Manager for review of the inclusion and exclusion criteria, a potential subject's attending physician will be contacted to review the patient's study eligibility. If the attending is in agreement with the information collected by the UPMC Health Plan Case Manager, the patient will be eligible to be consented by the Research Assistant.

The Research Assistant will then approach the patient to explain the entire research project and obtain written and oral informed consent. Once informed consent is obtained, an enrollment questionnaire will be completed, which consists of the following components: 1) Medication adherence using the MMAS-4 (Morisky 4-Item Self-Report Measure of Medication-Taking Behavior) and CRN-2 (Cost-related non-adherence); 2) Cognitive status assessment using the MMSE; 3) Delirium assessment using the CAM; 4) EMMA Medication Delivery Unit proficiency testing; 5) Demographics and appointment scheduling. If the patient does not meet any of the additional exclusion criteria contained within the enrollment questionnaire, the patient will be considered to be enrolled in the study.

Randomization process: Subjects meeting all inclusion and exclusion criteria will randomized based on the number of medications that are prescribed: > 5 medications (polypharmacy group) or < 5 medications (non-polypharmacy group). Once a determination that a patient is in the polypharmacy or non-polypharmacy group, the research assistant will select a sequentially numbered envelope from either the polypharmacy or non-polypharmacy envelope stack. The envelope will contain a randomization sequence number that determines if the patient will be enrolled in the control or intervention group.

Discharge Planning and Transitional Care Control group: For those enrolled in the intervention group, the UPMC Health Plan will work with RxPartners LTC (wholly owned subsidiary of UPMC) to perform a medication regimen review and complete a "cost out" for patients who are expected to leave within 24 hrs. For those enrolled in the control group, the patient will be discharged from the hospital, but get their medications dispensed through RXPartners in traditional pill bottles. They will then continue to manage their medications in the same way that they had been prior to the study which may include taking medications directly from pill bottles or from a pill-box/reminder system.

Intervention group: For those enrolled in the intervention group, the UPMC Health Plan will work with RxPartners LTC (wholly owned subsidiary of UPMC) to perform a medication regimen review and complete a "cost out" for patients who are expected to leave within 24 hrs. The medication regimen review ensures that the currently prescribed medications are available to RxPartners and can be loaded and dispensed in the EMMA medication delivery unit (MDU). Only solid form medications of a certain size and shape can be packaged in the required blister-packs. The cost out procedure ensures that the insurance company will allow a medication to be filled potentially before the usual refill date (i.e., obtain a new prescription for a previously prescribed medication that already has an existing supply). We will also determine if the research study has funds sufficient to cover the federally-mandated collection of co-pays for newly dispensed medications. If the medication regimen review is deemed appropriate AND there are sufficient research resources to pay the patient's co-pay, then the patient will be retained in the study. The patient will then be asked to complete the EMMA Enrollment Questionnaire to ensure proper communication and scheduling of medication drops based on the patient's preferences. Finally, the patient will complete the Emed appointment information and reminder sheet to ensure appropriate in-home follow-up following discharge.

As part of the previously established medication reconciliation process in use at Presbyterian Hospital, the final medication list will be faxed to RxPartner's secure fax server. RxPartners will then dispense, blister pack, load an EMMA medication delivery unit, and print patient-specific medication information. Once all medications have been loaded, RxPartners will use their existing courier system to deliver the EMMA MDU and the patient-specific medication information directly to the patient's home M-F, located in a predefined geographic radius within 6 hours. RxPartners will also set up the EMMA MDU in the patient's home, and ensure that it can communicate with the INRange Systems server using its built-in wireless modem. If it cannot connect for whatever reason, the machine can be plugged directly into an analog phone line, previously determined to be present.

In summary, all medications being used in this project are medications that have been prescribed for clinical care by the patients' attending physicians. The only research portions are the use of the EMMA MDU and the specific research assessments described in this proposal. All other aspects of this proposal are being done for clinical care.

Follow-up Procedures:

Within 72 hours of hospital discharge, an EMS Care Transition Coach will visit all patients (regardless of control or intervention assignment) in their home based on their time preference. The primary goal of the home visit is to reconcile all of the patient's medication regimens (e.g., pre-hospitalization and post-hospitalization medications, over-the- counter medications, and medications prescribed to someone else that the patient is taking).

The Medication Discrepancy Tool will be used between the research team members to communicate possible problems but will not be given to the patient. For each potential medication discrepancy, we will directly contact and clarify the medication regimen with the patient's primary care provider (PCP) or Cardiologist. The coach will also confirm that the patient will be seen by his or her PCP within 7 days.

Additional follow-up procedures for the control and intervention group are detailed below:

Control group: An EMS Care Transition Coach will perform medication adherence and safety assessments, as well as home-based prevention and disease management for common cardiac conditions. Medication adherence will be determined in the control groups at days 1 (along with medication reconciliation), 45 and 90 (along with the exit-interview) through the use of a manual pill count procedure. If significant medication safety issues are noted during the day 45 visit, including improper storage, labeling, administration, and non-compliance to entire medication regimen, the UPMC Health Plan Case Manager will be contacted to potentially intervene. At the day 45 visit, the EMS Care Transition Coach will also conduct home-based prevention and disease management for common cardiac conditions using materials developed by the American Heart Association (AHA) Answers by Heart Fact Sheets.

Intervention group: At the day 45 visit, the EMS Care Transition Coach will conduct home-based prevention and disease management for common cardiac conditions using materials developed by the American Heart Association (AHA) Answers by Heart Fact Sheets.

Additionally, throughout the study the EMMA MDU has the ability to detect medication adherence in real-time. Therefore, we will program that the EMMA MDU generate an alert email to the UPMC Health Plan Case Manager who will be assigned to the patient upon discharge. This is a different UPMC Case Manager then the one that might have seen the patient in the hospital setting. Case managers are typically assigned to high-risk patients, such as those that we have enrolled with medication adherence problems. We will operationalize medication non-adherence as follows: 1) <80% overall medication adherence OR 2) >/= 2 missed doses of the same medication.

During the course of the study, if a new medication is needed, RxPartners will be responsible for blister-packing the medication (in the intervention group) or dispensing in traditional pill bottles, and either couriering it to the patient within 6 hours or delivering non-urgent medications through overnight-mail.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years of age.
2. Admitted during the study period for a nonpsychiatric condition to UPMC Presbyterian Hospital.
3. Documented in their medical record with a common cardiac condition.
4. Prescribed > 3 and < 20 regularly scheduled (i.e., non-PRN) prescription medications.
5. Be from and return to a home setting (not to an assisted living or skilled nursing facility, or to a program for all-inclusive care of the elderly, etc).
6. Reside within a predefined geographic radius of the hospital (specifically, Allegheny, Beaver, Butler, Fayette, Washington or Westmoreland Counties).
7. Have a working telephone.
8. Be English-speaking.
9. Have an informal caregiver or support person.
10. Evidence of unintentional medication non-adherence

Exclusion Criteria:

1. Have an active prescription for narcotic analgesic.
2. Enrolled in or plan to enroll into hospice care.
3. Plans to travel during the next 90 days following discharge for >/= 14 consecutive days.
4. Participating in another research protocol.
5. Have evidence in the chart of a diagnosis of active delirium.
6. Have evidence in the chart of a diagnosis of dementia.
7. Have evidence in the chart of legal blindness.
8. Unable to demonstrate appropriate use of the EMMA medication delivery unit.
9. Unable to receive ATT wireless service data plan based on physical address.
10. Evidence of intentional medication non-adherence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-05; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M. Handler, MD, PhD, CMD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Presbyterian Hospitl, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the study period, between May 15, 2012 and March 1, 2013, potentially eligible subjects were recruited at UPMC Presbyterian and UPMC Passavant Hospitals. Study eligibility was determined by electronic medical record review and bedside assessment.
Period: Overall Study
Arm/Group | Computerized Medication Delivery Unit | Usual Care
Started | 7 | 4
Completed | 7 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Computerized Medication Delivery Unit | Usual Care | Total
Number analyzed (Participants) | 7 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (12.4) | 71.1 (13.5) | 68.0 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence
Description: Will be measured by: (number of doses/ doses scheduled; EMMA (intervention) vs. determined by manual monthly pill counts (control))
Time Frame: 90-day
Measure: Mean (Standard Deviation); unit: percentage of medication adherence
Arm/Group | Computerized Medication Delivery Unit | Usual Care
Number analyzed (Participants) | 7 | 4
percentage of medication adherence | 97.5 (3.9) | 87.2 (15.0)

2. Secondary Outcome: Medication-reconciliation Errors During Transition From Hospital to Home
Description: Using the previously validated and reliable medication discrepancy tool (MDT)
Time Frame: 90-day
Measure: Number; unit: Participants with errors
Arm/Group | Computerized Medication Delivery Unit | Usual Care
Number analyzed (Participants) | 7 | 4
Participants with errors | 0 | 0

3. Secondary Outcome: Hospital Readmission Rates
Description: Determine the percentage of patients that are readmitted to the hospital within 30 days of discharge
Time Frame: 30 day
Measure: Number; unit: % readmissions
Arm/Group | Computerized Medication Delivery Unit | Usual Care
Number analyzed (Participants) | 7 | 4
% readmissions | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the 90 day duration of the study.
Arm/Group | Computerized Medication Delivery Unit | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/4
Other Adverse Events (participants affected / at risk) | 0/7 | 0/4

LIMITATIONS AND CAVEATS:
We terminated the study early after exhausting all possible approaches to increasing participant enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No